CLINICAL TRIAL: NCT07258953
Title: The Effects of Intramuscular Injection Using ShotBlocker, Cold Needling, and Both Methods in Combination on Pain and Satisfaction: A Randomized Controlled Trial
Brief Title: ShotBlocker, Cold Needling, and Both Methods in Combination Pain and Satisfaction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Yadigar Ordu, Associate Professor, Necmettin Erbakan University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: ShotBlocker and Cold Needle
Record Dates: First submitted 2025-09-26; First posted 2025-12-02 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: Group 1: ShotBlocker Group 2: Cold Needle Group 3: ShotBlocker + Cold Needle Group 4: Control
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Patients will be randomly assigned to groups and each will be taken individually to the injection unit.
  All injections will be administered by a single nurse working in the unit where the injections will be administered. The researcher will participate solely as an observer, will not intervene, and will not know which patient is in which group.
  Data obtained from the study will be coded as A, B, C, and D and submitted for statistical analysis.
  By concealing the group information, the analysis will be conducted objectively.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ShotBlocker+cold needle (Experimental): During intramuscular injection, ShotBlocker and the cold needle will be used simultaneously.
  Interventions: Other: ShotBlocker+cold needle
- Cold needle (Experimental): ShotBlocker will be used during intramuscular injection.
  Interventions: Other: ShotBlokcer
- ShotBlocker (Experimental): A cold needle will be used during intramuscular injection.
  Interventions: Other: Cold needle
- Control (Placebo Comparator): Intramuscular injections will be performed according to standard technique.
  Interventions: Other: Control

INTERVENTIONS:
Other: ShotBlocker+cold needle — During intramuscular injection, ShotBlocker and the cold needle will be used simultaneously.
  Arms: ShotBlocker+cold needle
Other: Cold needle — A cold needle will be used during intramuscular injection.
  Arms: ShotBlocker
Other: ShotBlokcer — ShotBlocker will be used during intramuscular injection.
  Arms: Cold needle
Other: Control — Intramuscular injection will be conducted according to standard technique.
  Arms: Control

SUMMARY:
Intramuscular (IM) injections are one of the most frequently used pharmacological treatment methods in nursing practice. Reducing the pain experienced by patients during this procedure and ensuring patient satisfaction are important indicators of treatment quality. Reducing injection-related pain should be a priority in nursing care for both patient safety and the effectiveness of the treatment process.

This study is a triple-blind, randomized, controlled trial. It was designed to evaluate the effects of ShotBlocker, cold needle, and a combination of both methods during intramuscular injection on patient pain levels and satisfaction. The research will be conducted in the injection unit affiliated with the Adult Emergency Department of Konya City Hospital, Ministry of Health of the Republic of Turkey. The study population will consist of patients who presented for cyanocobalamin injections, and the sample will consist of 132 individuals who voluntarily agreed to participate in the study and met the inclusion criteria. Before conducting the study, ethical approval will be obtained from the Necmettin Erbakan University Health Sciences Ethics Committee and from the Konya City Hospital of the Ministry of Health of the Republic of Turkey. Collected data will be analyzed using the SPSS statistical package program (version 22.0; SPSS Inc., USA). The Kolmogorov-Smirnov test will be used to assess whether the data exhibit a normal distribution; statistical significance will be accepted as p<0.05.

DETAILED DESCRIPTION:
In parallel with the changes and developments in the healthcare field worldwide and in Türkiye, it is crucial that nursing practices are based on scientific knowledge and are evidence-based. Nurses must integrate the most up-to-date information into their practices in patient care. Medication administration, a fundamental element of medical treatment, is among nurses' legal responsibilities and requires great professional care and meticulousness. Medication administration is performed by nurses through various routes, including parenteral, topical, inhalation, and oral administration.

Intramuscular injection is a parenteral drug administration method, administering the medication deep into muscle tissue. It is frequently used in clinical practice. It is a riskier procedure than other injection methods, so it should be performed by professionals.

Intramuscular injections can lead to serious complications if the correct technique is not used. These complications include nerve damage, vascular or tissue damage, infection, abscess, hematoma, tissue necrosis, muscle stiffness, tingling, and the rare Nicolau syndrome. The most common complication is pain during the injection. In one study, participants underwent intravenous, intramuscular, and spinal injections, and when pain levels were compared, it was determined that the highest pain level was felt during the intramuscular injection. This result suggests that intramuscular injections may cause more pain compared to other injection types. Reducing the pain felt due to needle insertion during intramuscular injection alleviates individuals' anxiety and fears about the procedure and contributes to an increase in their satisfaction with the injection procedure. There are studies on the level of satisfaction with intramuscular injection procedures. These are: Techniques such as acupressure , ShotBlocker , cold needling , helfer skin tap (HSTT) , and vibration stimulation have been found to increase patient satisfaction with the treatment. Pharmacological, non-pharmacological, and surgical techniques can be used to reduce pain. Firstly, the use of non-pharmacological methods to control pain is important. Accordingly, nurses utilize various nonpharmacological methods to reduce pain and increase patient comfort. Correct patient positioning, use of appropriate equipment, changing the needle tip after withdrawal, and applying the Z technique and the airlock technique for irritating medications are effective in reducing pain during intramuscular injections. Additionally, skin stimulation techniques such as massage, menthol application, ShotBlocker, vibration, hot-cold application, cold needle technique, Buzzy, TENS, manual pressure, and helfer skin tap, as well as cognitive methods such as listening to music, relaxation, and distraction are also helpful in relieving pain. According to Gate Control Theory, one of the theories used to reduce pain, mechanical stimuli such as touch or manual pressure activate large nerve fibers, blocking the pain signals carried by small fibers in the spinal cord. This prevents the brain from perceiving the pain signal. Manual pressure applied before the injection allows the release of natural pain-relieving hormones such as endorphins, which raises the pain threshold. It increases blood circulation, reduces the perception of pain, and promotes tissue healing. Thanks to these mechanisms, pain can be effectively reduced through non-pharmacological methods. Literature has shown that the helfer skin tap technique reduces pain in newborns, children, and adults. Internal rotation of the extremity during intramuscular injection has been found to be effective in reducing injection pain and relaxing muscles. Various clinical studies in different age groups have shown that Buzzy is effective in reducing pain during needle procedures. The ShotBlocker, with its ridged surface applied by pressing on the skin, helps reduce the perception of pain by providing a physical stimulus with its blunt tips during injection. Its mechanism of action is that the projections exert pressure on the skin by stimulating fast nerve endings, temporarily blocking slower pain signals. This method reduces pain. Studies on children and adults have found it effective in reducing pain. Studies on the use of cold application and cold spray have determined that these methods significantly reduce post-injection pain. Studies using the cold needle technique show that this method is effective in reducing pain felt during injections in both children and adults. This technique is implemented by cooling the syringe tip to 0-2°C before injection and aims to reduce the patient's perception of pain during the injection. A review of the literature reveals that many studies have been conducted using various methods to reduce pain during intramuscular injection. Studies comparing ShotBlocker with other methods are quite common. However, the number of studies on the cold needle technique is limited. Only one study has been found in the literature that evaluated the effects of ShotBlocker and cold needle methods on pain and satisfaction during injection.

This study is the first to compare the effects of ShotBlocker and cold needle methods on pain and satisfaction during intramuscular injection, and to examine the effects of using these two methods together on pain and satisfaction during intramuscular injection. The lack of any studies in the literature on the simultaneous use of these two methods makes this study scientifically original. In this context, the study will not only make an innovative contribution to existing knowledge but also have the potential to develop concrete and applicable solutions to increase patient satisfaction in nursing practice. It is believed that the data obtained regarding the combined use of these easy-to-implement, economical, and time-practical methods will make unique contributions to both clinical practice and the literature.

ELIGIBILITY:
Inclusion Criteria:

1. Must be between 18 and 65 years of age.
2. Must have no problems speaking and understanding Turkish.
3. Must have been prescribed 1000 mcg (1 ml ampoule) of cyanocobalamin IM injection.
4. Must use the deltoid region for the injection.
5. Must not be in the menstrual cycle.
6. Must not be pregnant.
7. Must have no history of diabetes.
8. Must have a Body Mass Index (BMI) between 18.5 and 30.
9. Must have no scars, incisions, lipodystrophy, or infection at the injection site.
10. Must have no history of allergy to the medication.
11. Must have no pain, fear, etc. The inclusion criteria for the study were: not having any illness that prevents the perception of variables (vision, hearing, sensory loss, cognitive impairment, stroke, etc.),
12. not using centrally or peripherally acting analgesics or sedatives,
13. not having limb impairments,
14. having a VAS score of "0" before the injection,
15. agreeing to participate in the study.

Exclusion Criteria:

1. Chronic or acute pain,
2. Receiving oral or parenteral analgesic treatment before the study,
3. Receiving another injection in the deltoid region,
4. Developing a drug-related allergy or other complication,
5. Having a contact-related infectious disease,
6. Participants wishing to withdraw from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2026-01-01 (Actual); Primary Completion 2026-04-10 (Estimated); Study Completion 2026-06-10 (Estimated)

PRIMARY OUTCOMES:
Visual Pain Scale (VAS) | up to 5 months
  After the injection, the pain level will be determined using VAS.The lowest VAS score is "0" and the highest is "10." A higher score indicates greater pain.

SECONDARY OUTCOMES:
Injection satisfaction | up to 5 months
  After the injection, patient satisfaction will be assessed. At this stage, patients will be asked to rate their satisfaction on a scale of 1-10.

CONTACTS AND LOCATIONS:
Overall Officials: Yadigar Yadigar, Principal Investigator — Necmettin Erbakan University
Locations (1):
- Necmettin Erbakan University, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No